CLINICAL TRIAL: NCT00006347
Title: Phase I Non-Myeloablative Trial With 90Y-Humanized MN-14 (Anti-CEA) Antibody for Relapsed or Refractory Small Cell Lung Cancer (SCLC)
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Relapsed or Refractory Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068199; CMMI-C-057A-99; NCI-H00-0064
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2003-04

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Indium

INTERVENTIONS:
Radiation: indium In 111 monoclonal antibody MN-14
Radiation: yttrium Y 90 monoclonal antibody MN-14

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have relapsed or refractory small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose limiting toxicity and maximum tolerated dose of yttrium Y 90 anti-CEA monoclonal antibody MN-14 in patients with relapsed or refractory small cell lung cancer.
* Determine the dosimetric and pharmacokinetic properties of this treatment regimen in the blood, normal organs, and tumors of these patients.
* Determine the stability and complexation with circulating carcinoembryonic antigen of this radioantibody in the plasma of these patients.
* Determine the antibody response of these patients treated with this regimen.
* Determine the antitumor effects of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study of yttrium Y 90 anti-CEA monoclonal antibody MN-14 (90Y-hMN-14). Patients are stratified according to prior radiotherapy (yes vs no).

Patients undergo pretherapy imaging with indium In 111 anti-CEA monoclonal antibody MN-14 IV over 30-40 minutes on day -7 or -6 followed by external scintigraphy on days -7 or -6 to 0.

Patients who show positive localization of at least one documented tumor site receive 90Y-hMN-14 IV over 30-40 minutes on day 0.

Cohorts of 3-6 patients receive escalating doses of 90Y-hMN-14 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

Patients are followed at 2, 4, 8, and 12 weeks; every 3 months for 2 years; and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 10-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)

  * Must have received at least one prior course of standard chemotherapy and, if indicated, up to 6,900 cGy of thoracic radiotherapy
  * Patients who received prior radiotherapy must show evidence of progressive disease
  * Patients who received no prior radiotherapy to the primary tumor must show evidence of stable or progressive disease
* Measurable disease
* Must have evidence of carcinoembryonic antigen (CEA) production or expression documented by one of the following:

  * Serum CEA at least 10 ng/mL
  * Positive immunohistology of either the primary tumor or a metastasis with CEA specific monoclonal antibody
* Must have unilateral bone marrow biopsy with less than 25% tumor involvement
* No known, active brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%
* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 mg/dL
* AST no greater than 2 times upper limit of normal (ULN)
* No hepatitis B or C
* No other serious liver abnormality

Renal:

* Creatinine no greater than 1.5 times ULN
* No urinary incontinence

Cardiovascular:

* Ejection fraction at least 50%

Pulmonary:

* FEV_1 and FVC at least 60%
* DLCO at least 50% predicted

Other:

* No severe anorexia, nausea, or vomiting
* No other significant medical problems
* No prisoners
* No reactivity to humanized MN-14 (in patients with prior exposure to chimeric or humanized antibody)
* HIV negative
* No active HIV-related disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months following study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* No concurrent growth factors (e.g., filgrastim [G-CSF])

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No prior high dose chemotherapy with stem cell transplantation

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* Prior radiotherapy to less than 30% of red marrow (including standard chest x-ray for limited stage SCLC) allowed

Surgery:

* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (1):
- Garden State Cancer Center, Belleville, New Jersey, United States